CLINICAL TRIAL: NCT03176797
Title: Quantitative Diagnosis of Liver Fibrosis on Multiparametric MRI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Quan Xianyue, Professor, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LC2016PY034
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Liver Fibrosis; Cirrhosis
Keywords: Liver Fibrosis, multiparametric magnetic resonance imaging
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver MRI (Experimental): Liver MRI including DWI, IVIM, DKI, T1ρ, T1 mapping of pre-contrast and hepatocyte phase and SWI.
  Interventions: Diagnostic Test: Liver MRI

INTERVENTIONS:
Diagnostic Test: Liver MRI — Liver MRI including DWI, IVIM, DKI, T1ρ, T1 mapping of pre-contrast and hepatocyte phase and SWI.

SUMMARY:
Early diagnosis and treatment of liver fibrosis can repress or delay the development of cirrhosis and hepatocellular carcinoma. The purpose of this pilot study is to evaluate non-invasive multiparametric magnetic resonance imaging (MRI) techniques in the detection and grading of liver fibrosis, so that patients can be treated in time. These techniques combined could reach high diagnostic performance for detection of liver fibrosis, and could decrease the number of liver biopsies.

DETAILED DESCRIPTION:
Early diagnosis and treatment of liver fibrosis can repress or delay the development of cirrhosis and hepatocellular carcinoma. While liver biopsy is still considered the gold standard for diagnosing and assessing the presence and degree of liver fibrosis and inflammation, it has disadvantages including the potential for sampling error and risk of complications. New imaging modalities such as diffusion weighted imaging (DWI), intravoxel incoherent motion (IVIM), diffusion kurtosis imaging (DKI), T1ρ relaxation time (T1ρ), T1 mapping of pre-contrast and hepatocyte phase using hepatocyte specific agent and susceptibility weighted imaging (SWI) allow non-invasive evaluation of liver parenchymal characteristics and may be able to detect and quantify parenchymal fibrosis alleviating the need for biopsy. Patients with chronic liver disease or normal liver parenchyma who are scheduled to undergo either liver resection or liver biopsy are included. Referred patients undergo multiparametric MRI including DWI, IVIM, DKI, T1ρ, T1 mapping of pre-contrast and hepatocyte phase and SWI before surgery or biopsy. The pathologic changes are evaluated using multiparametric MRI, and compared between normal/early fibrosis and advanced fibrosis. To explore if combine these techniques could reach higher diagnostic performance for detection and grading of liver fibrosis. This project will provide a reliable and noninvasive method for the monitoring stage of liver fibrosis and therapeutic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* chronic liver disease (viral hepatitis, alcoholic hepatitis, or other...)
* AND willingly able to complete all research procedures and follow the entire research process
* AND scheduled for liver resection or biopsy
* AND signed informed consent

Exclusion Criteria:

* Any contraindication for contrast-enhanced MRI
* Pregnant or nursing women
* Any organ transplant history, and existing functional grafts (except corneal or fur grafts)
* Recent right upper quadrant patients with traumatic healed
* A serious history of illness or other evidence of a serious illness or suffering from any other disease
* Patients who have been enrolled in other interventional clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI T1ρ T1mapping SWI and DWI | MRI within 3 months of liver biopsy or surgery
  Quantitative Diagnosis accuracy of MRI in the degree of fibrosis and advanced fibrosis compared with histology

SECONDARY OUTCOMES:
MRI T1ρ T1mapping SWI and DWI | Blood Test taken on same day as MRI
  Quantitative Diagnosis accuracy of MRI in the degree of fibrosis and advanced fibrosis compared with serological markers.

CONTACTS AND LOCATIONS:
Overall Officials: Xianyue Quan, MD, Principal Investigator — Southern Medical University, China
Locations (1):
- ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kobayashi K, Nakao H, Nishiyama T, Lin Y, Kikuchi S, Kobayashi Y, Yamamoto T, Ishii N, Ohashi T, Satoh K, Nakade Y, Ito K, Yoneda M. Diagnostic accuracy of real-time tissue elastography for the staging of liver fibrosis: a meta-analysis. Eur Radiol. 2015 Jan;25(1):230-8. doi: 10.1007/s00330-014-3364-x. Epub 2014 Aug 23. PMID 25149296
- [Result] Friedrich-Rust M, Rosenberg W, Parkes J, Herrmann E, Zeuzem S, Sarrazin C. Comparison of ELF, FibroTest and FibroScan for the non-invasive assessment of liver fibrosis. BMC Gastroenterol. 2010 Sep 9;10:103. doi: 10.1186/1471-230X-10-103. PMID 20828377
- [Result] Wang YX, Yuan J, Chu ES, Go MY, Huang H, Ahuja AT, Sung JJ, Yu J. T1rho MR imaging is sensitive to evaluate liver fibrosis: an experimental study in a rat biliary duct ligation model. Radiology. 2011 Jun;259(3):712-9. doi: 10.1148/radiol.11101638. Epub 2011 Mar 24. PMID 21436087
- [Result] Zhao F, Wang YX, Yuan J, Deng M, Wong HL, Chu ES, Go MY, Teng GJ, Ahuja AT, Yu J. MR T1rho as an imaging biomarker for monitoring liver injury progression and regression: an experimental study in rats with carbon tetrachloride intoxication. Eur Radiol. 2012 Aug;22(8):1709-16. doi: 10.1007/s00330-012-2419-0. Epub 2012 Mar 27. PMID 22752522
- [Result] Girometti R, Furlan A, Esposito G, Bazzocchi M, Como G, Soldano F, Isola M, Toniutto P, Zuiani C. Relevance of b-values in evaluating liver fibrosis: a study in healthy and cirrhotic subjects using two single-shot spin-echo echo-planar diffusion-weighted sequences. J Magn Reson Imaging. 2008 Aug;28(2):411-9. doi: 10.1002/jmri.21461. PMID 18666139
- [Result] Hu G, Chan Q, Quan X, Zhang X, Li Y, Zhong X, Lin X. Intravoxel incoherent motion MRI evaluation for the staging of liver fibrosis in a rat model. J Magn Reson Imaging. 2015 Aug;42(2):331-9. doi: 10.1002/jmri.24796. Epub 2014 Nov 11. PMID 25384923
- [Result] Shiha G, Ibrahim A, Helmy A, Sarin SK, Omata M, Kumar A, Bernstien D, Maruyama H, Saraswat V, Chawla Y, Hamid S, Abbas Z, Bedossa P, Sakhuja P, Elmahatab M, Lim SG, Lesmana L, Sollano J, Jia JD, Abbas B, Omar A, Sharma B, Payawal D, Abdallah A, Serwah A, Hamed A, Elsayed A, AbdelMaqsod A, Hassanein T, Ihab A, GHaziuan H, Zein N, Kumar M. Asian-Pacific Association for the Study of the Liver (APASL) consensus guidelines on invasive and non-invasive assessment of hepatic fibrosis: a 2016 update. Hepatol Int. 2017 Jan;11(1):1-30. doi: 10.1007/s12072-016-9760-3. Epub 2016 Oct 6. PMID 27714681
- [Result] Petitclerc L, Sebastiani G, Gilbert G, Cloutier G, Tang A. Liver fibrosis: Review of current imaging and MRI quantification techniques. J Magn Reson Imaging. 2017 May;45(5):1276-1295. doi: 10.1002/jmri.25550. Epub 2016 Dec 16. PMID 27981751
- [Result] Hu G, Zhang X, Liang W, Zhong X, Chan Q, Lin X, Lin T, Li Y, Quan X. Assessment of liver fibrosis in rats by MRI with apparent diffusion coefficient and T1 relaxation time in the rotating frame. J Magn Reson Imaging. 2016 May;43(5):1082-9. doi: 10.1002/jmri.25084. Epub 2015 Oct 26. PMID 26497954